CLINICAL TRIAL: NCT04971291
Title: A Randomized, Active-Controlled, Evaluation of AXS-05 for the Treatment of Treatment Resistant Depression in Treatment-Adherent Patients
Brief Title: An Evaluation of AXS-05 for the Treatment of TRD in Treatment-Adherent Patients
Acronym: TARGET
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AXS-05-TRD-203
Record Dates: First submitted 2021-07-12; First posted 2021-07-21 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Major Depressive Disorder; Treatment Resistant Depression
Keywords: AXS-05; Axsome; NMDA receptor
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AXS-05 (Experimental): 45 mg dextromethorphan-105 mg bupropion
  Interventions: Drug: AXS-05
- Bupropion SR (Active Comparator): 150 mg bupropion
  Interventions: Drug: Bupropion SR

INTERVENTIONS:
Drug: AXS-05 — AXS-05 taken twice daily for 6 weeks
  Arms: AXS-05
Drug: Bupropion SR — Bupropion taken twice daily for 6 weeks
  Arms: Bupropion SR

SUMMARY:
The TARGET study is an active-controlled evaluation of AXS-05 compared to bupropion in patients with treatment-resistant major depressive disorder (MDD) who are adherent to study drug. Subjects are considered to have treatment-resistant MDD if they have had a historical inadequate response to 1 or 2 prior antidepressant treatments (ADTs) and a prospective inadequate response to treatment with bupropion SR, during the current major depressive episode.

The TARGET study will first determine treatment adherence based on analysis of drug concentrations of dextromethorphan (in the AXS-05 group) and bupropion (in the bupropion group), and then evaluate the efficacy of AXS-05 in patients determined to be treatment-adherent. Efficacy data for evaluation of treatment effect will be obtained from assessments made during study AXS-05-301.

ELIGIBILITY:
Key Inclusion Criteria:

* Provided written informed consent to participate in Study AXS-05-301
* Has treatment-resistant depression, defined as an inadequate response to 2 or 3 prior ADTs
* Body mass index (BMI) between 18 and 40 kg/m2, inclusive

Key Exclusion Criteria:

* Suicide risk
* Treatment with any investigational drug within 6 months
* History of electroconvulsive therapy (ECT), vagus nerve stimulation, transcranial magnetic stimulation, or any experimental central nervous system treatment during the current episode or in the past 6 months
* Pregnant, breastfeeding, or planning to become pregnant or breastfeed during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2021-04-14 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) total score | Change from Baseline to Week 6
  The MADRS is used to assess depressive symptomatology during the previous week. Subjects are rated on 10 items to assess feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating and lack of interest. Each item is scored on a 7-point scale. A score of 0 indicates the absence of symptoms, and a score of 6 indicates symptoms of maximum severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Axsome Research Site, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No